CLINICAL TRIAL: NCT07295457
Title: Randomized Clinical Trial Evaluating the Efficacy and Implementation of an Early Adapted Physical Activity to Prevent and Manage Aromatase Inhibitor-induced Musculoskeletal Pain in Breast Cancer
Brief Title: Clinical Trial Evaluating the Efficacy and Implementation of an Early Adapted Physical Activity to Prevent and Manage Aromatase Inhibitor-induced Musculoskeletal Pain in Breast Cancer (APIS)
Acronym: APIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL24_0748
Record Dates: First submitted 2025-09-26; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Hormonotherapy; Musculoskeletal pain; Adapted physical activity; Aromatase inhibitors; Exercise oncology; Implementation science
MeSH Terms: conditions — Breast Neoplasms; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: The APIS study is a hybrid Type 1 Effectiveness-Implementation randomized clinical trial that combines the evaluation of:
  * The effectiveness of an APA program on AIMSS : multicenter, controlled, randomized, 2-parallel group, open-label, prospective, minimal risk and constraint interventional clinical research study.
  * Implementation, exploring, using the RE-AIM (Reach Effectiveness Adoption Implementation Maintenance) theoretical framework, its adoption, accessibility, practical integration into care pathways, and sustainability in different settings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted Physical Activity started early (announcement) (Experimental): The APA (Adapted Physical Activity) program is decided during the initial assessment.
  Interventions: Behavioral: Adapted Physical Activity started early
- Adapted Physical Activity begins at the start of hormone therapy (control group). (Active Comparator): Patients will receive standard care. The personalized APA (Adapted Physical Activity) protocol will begin at the same time as hormone therapy. Hormone therapy is initiated at the end of primary treatment and continues during the survivorship care period.
  Interventions: Behavioral: Adapted Physical Activity begins at the start of hormone therapy

INTERVENTIONS:
Behavioral: Adapted Physical Activity started early — The Adapted Physical Activity program is decided during the initial assessment. The total duration of the rehabilitation protocol is 12 weeks, with 2 one-hour sessions per week.
  The rehabilitation protocol chosen in this study is mixed, i.e. it combines :
  * Exercise training on ergocyclometer or treadmill
  * Flexibility and muscle-strengthening work supervised by a physiotherapist
  * Free work with the APA practitioner
  Arms: Adapted Physical Activity started early (announcement)
Behavioral: Adapted Physical Activity begins at the start of hormone therapy — Adapted Physical Activity begins at the start of hormone therapy The total duration of the rehabilitation protocol is 12 weeks, with 2 one-hour sessions per week.
  The rehabilitation protocol chosen in this study is mixed, i.e. it combines :
  * Exercise training on ergocyclometer or treadmill
  * Flexibility and muscle-strengthening work supervised by a physiotherapist
  * Free work with the APA practitioner
  Arms: Adapted Physical Activity begins at the start of hormone therapy (control group).

SUMMARY:
Aromatase inhibitors (AI) are the standard adjuvant hormone therapy for postmenopausal women with hormone-sensitive breast cancer. However, nearly half of patients experience AI-induced musculoskeletal symptoms (AIMSS), particularly pain, which compromise quality of life and treatment adherence. While adapted physical activity offers proven benefits in oncology, its specific role in preventing or managing AIMSS remains unclear. Moreover, the maintenance of physical activity during the care pathway in real-world settings is limited, highlighting the need for hybrid approaches that evaluate both clinical effectiveness and implementation. In response to these challenges, the primary study aim will be to compare the prevalence of musculoskeletal pain after six months of aromatase inhibitor therapy between patients initiating a personalized adapted physical activity program at the beginning of the care pathway and those receiving usual care. Secondary aims will be to (1) assess additional effects of the intervention on physical health, psychosocial well-being and treatment adherence, (2) explore contextual factors influencing program implementation in routine oncology care and (3) identify potential risk factors for the development of AIMSS. The APIS study is a hybrid type I effectiveness-implementation randomized controlled trial including 182 postmenopausal women with non-metastatic hormone-sensitive breast cancer. APIS will generate new evidence on the clinical and implementation effectiveness of early personalized APA (Adapted Physical Activity) in preventing AIMSS. The hybrid design will support the development of sustainable, patient-centered interventions, potentially improving quality of life, adherence to AI therapy and long-term outcomes in breast cancer survivorship.

Ancillary study (Groupement Hospitalier Nord, Hospices Civils de Lyon) The humero-scapulo-thoracic region is particularly exposed to functional alterations during the course of care of patients treated for breast cancer. In addition to the loss of strength and mobility associated with surgical and medical treatment, the shoulder can also be the site of pain due to AIMSS or PMDS (Post-Mastectomy Pain Syndrome).

These pains are often studied separately, depending on the treatment, but few studies offer a global vision of the functional evolution of the shoulder throughout the course of care, enabling prevention and adjustment of management. It is also relevant to assume that early APA treatment could improve functional rehabilitation in this area.

The aim of this study is therefore to evaluate the impact of an APA assessment and early referral to a personalized program (APIS protocol) on shoulder functionality, depending on the time of intervention in the therapeutic pathway.

ELIGIBILITY:
Inclusion Criteria:

Quantitative study:

* Women aged 18 to 75
* Person with non-metastatic breast cancer
* positive for at least one hormone receptor
* Person treated with an Aromatase Inhibitor
* Person with the following treatment regimen: Surgery - radiotherapy - aromatase inhibitor hormone therapy or surgery - chemotherapy (neoadjuvant or adjuvant) +/- targeted therapy - radiotherapy - aromatase inhibitor hormone therapy.
* Person affiliated to a social security scheme
* Person having signed a free and informed consent

Qualitative study:

For patients :

* Patient having given consent to participate in the APIS study
* Patient agreeing to participate in the qualitative study (box checked on the APIS informed consent form)
* Patient agreeing to the recording of the semi-directive interview

For healthcare professionals :

* Person practicing within the Saint-Étienne University Hospital and the Croix-Rousse University Hospital as a surgeon, oncologist, radiotherapist, sports medicine physician, APA instructor, physiotherapist, head nurse, care coordinator nurse, or advanced practice nurse
* Persons working with patients treated with aromatase inhibitors for non-metastatic breast cancer
* Person who has received individual information
* Person who has given consent to participate in the study
* Person agreeing to the recording of the semi-directive interview
* Person of legal age

Ancillary study :

* Eligible patient who has given consent to participate in the APIS study
* Patient agreeing to participate in the ancillary study (box checked on the APIS informed consent form)

Exclusion Criteria:

For all patients:

* Person deprived of liberty by judicial or administrative decision
* Person under psychiatric care (unstable pathology)
* Person of full age under legal protection (guardianship, curatorship)
* Person unable to receive sufficient information due to impaired higher functions, or insufficient command of the French language
* Person participating in another interventional research study with an exclusion period still in progress at the time of pre-inclusion
* Person with absolute contraindications to physical exercise:

  * Unstable angina
  * Decompensated heart failure
  * Complex ventricular rhythm disorders
  * Uncontrolled severe arterial hypertension
  * Pulmonary arterial hypertension (> 60 mm Hg)
  * Presence of large or pedunculated intracavitary thrombus
  * Acute pericardial effusion
  * Severe obstructive cardiomyopathy
  * Tight and/or symptomatic aortic stenosis
  * Recent thrombophlebitis with or without pulmonary embolism
  * Diabetes with plantar perforator disease for physical activity activities involving the lower limbs
* Persons with musculoskeletal pathologies making cycling impossible

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Score of most intense musculoskeletal pain | 6 months after introduction of hormone therapy
  To analyze the impact of implementing a specific APA program, right from the start of treatment, on the prevalence of musculoskeletal pain experienced by patients treated for breast cancer with aromatase inhibitors (AI) after 6 months of hormone therapy (peak of symptoms).
  Musculoskeletal pain are measured using the Nordic-type questionnaire.
  This score is measured using the Nordic questionnaire, which includes a Numerical Rating Scale (NRS) for musculoskeletal pain ranging from 0 to 10:
  * 0 = no pain or discomfort
  * 10 = intolerable pain or discomfort A higher score reflects a more unfavorable clinical outcome.

SECONDARY OUTCOMES:
Evolution of musculoskeletal pain intensity | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Musculoskeletal pain is measuring using the evolution of the score of the Nordic Musculoskeletal Questionnaire. The score was compare between pre-therapy and 6 months of hormone therapy in experimental and control groups.
  The Nordic Musculoskeletal Questionnaire including a Numerical Rating Scale (range 0 - 10), with higher scores indicating more severe pain.
Score of global pain | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Global pain is measured using the numerical scale. The numerical scale is a self-assessment scale and consists of asking the patient to quantify her overall pain at the present moment on a virtual scale ranging from 0 (no pain) to 10 (maximum imaginable pain). The aim is to compare the effects of the intervention on overall health outcomes, including physical health and psychosocial well-being.
Evaluation of Quality of life | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Quality of life is measured using FACT-B (Functional Assessment of Cancer Therapy - Breast) scale associated with the endocrine subscale (ES).
  FACT-B scale is a validated instrument designed to assess health-related quality of life in patients with breast cancer. It includes 37 items covering five domains: physical well-being, social/family well-being, emotional well-being, functional well-being, and breast cancer-specific concerns. Each item is rated on a 5-point Likert scale ranging from 0 ("not at all") to 4 ("very much"). Scores are summed to yield a total FACT-B score ranging from 0 to 148, with higher scores indicating better quality of life.
  Endocrine subscale (ES) specifically assesses endocrine symptoms and includes 19 quantifiable items such as hot flushes, weight gain and joint pain. Items are scored using the same 0-4 Likert scale, resulting in a total ES score ranging from 0 to 76, with higher scores reflecting fewer endocrine symptoms and better quality of life.
Fatigue | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Fatigue is measured using FACIT Fatigue - version 4- (Functional Assessment of Chronic Illness Therapy - Fatigue) Scale. The aim is to compare the effects of the intervention on overall health outcomes, including physical health and psychosocial well-being.
  Patients respond using a 5-point Likert scale. Each response is scored from 0 ("not at all") to 4 ("very much").
  The scoring system reverses the numbers for negative items. This means that for 11 items with negative statements (such as "I feel tired"), a 4 becomes a 0 and a 3 becomes a 1. Adding the 13 scores gives a total between 0 and 52 points.
  Higher total scores mean less fatigue and a better quality of life. Scores below 30 indicate severe fatigue.
Anxiety | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Anxiety is measured using HAD (Hospital Anxiety and Depression) scale.The aim is to compare the effects of the intervention on overall health outcomes, including physical health and psychosocial well-being.
  The HAD scale is a tool used to screen for anxiety and depressive disorders. It consists of 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to depression (total D), thus yielding two scores (maximum score for each = 21).
  Interpretation:
  To screen for anxiety and depression symptoms, the following interpretation can be used for each score (A and D):
  * 7 or less: no symptoms
  * 8 to 10: possible symptoms
  * 11 or more: definite symptoms.
Cognitive complaints | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Cognitive complaints are measured using FACT-Cognitive Function -version 3 (Functional Assessment of Cancer Therapy - Cognitive Function) scale. The aim is to compare the effects of the intervention on overall health outcomes, including physical health and psychosocial well-being.
  The FACT-G comprises four subscales: physical well-being (PWB; 7 items, score range 0-28), social/family well-being (SWB; 7 items, score range 0-28), emotional well-being (EWB; 6 items, score range 0-24), and functional well-being (FWB; 7 items, score range 0-28).
  Negatively worded items are reverse-scored before summation, so that higher subscale and total scores indicate better self-reported cognitive functioning.
Physical condition | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Physical condition is measuring using the 6-minute walk test. The score (between 375 and 546) was compare between pre-therapy and 6 months of hormone therapy in experimental and control groups (higher score mean a better outcome).
Weight | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Body composition is assessed by weight (kg), height (cm), Body Mass Index (BMI = weight/height in meters squared), waist circumference, measurement of the four skinfolds (validated measurement for assessing adiposity: % body fat) and malnutrition screening (Malnutrition Universal Screening Tool - MUST).
  Weight is measured in kilograms
Height | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Body composition is assessed by weight (kg), height (cm), Body Mass Index (BMI = weight/height in meters squared), waist circumference, measurement of the four skinfolds (validated measurement for assessing adiposity: % body fat) and malnutrition screening (Malnutrition Universal Screening Tool - MUST).
  Height is measured in centimeters
Body Mass Index (BMI) | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Body composition is assessed by weight (kg), height (cm), Body Mass Index (BMI = weight/height in meters squared), waist circumference, measurement of the four skinfolds (validated measurement for assessing adiposity: % body fat) and malnutrition screening (Malnutrition Universal Screening Tool - MUST).
  Body Mass Index (BMI)
  * Description: BMI will be calculated by dividing weight (kg) by height (m)². Weight and height will be measured according to standardized procedures, but only BMI will be reported as an outcome measure, as these data are collected solely for its calculation.
  * Unit of measurement: kg/m²
  * Interpretation: Higher values reflect greater adiposity.
Waist circumference | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Body composition is assessed by weight (kg), height (cm), Body Mass Index (BMI = weight/height in meters squared), waist circumference, measurement of the four skinfolds (validated measurement for assessing adiposity: % body fat) and malnutrition screening (Malnutrition Universal Screening Tool - MUST).
  Waist circumference
  * Description: Waist circumference will be measured in centimeters.
  * Unit of measurement: cm
  * Interpretation: Higher values are associated with greater central adiposity.
Percentage of body fat | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Body composition is assessed by weight (kg), height (cm), Body Mass Index (BMI = weight/height in meters squared), waist circumference, measurement of the four skinfolds (validated measurement for assessing adiposity: % body fat) and malnutrition screening (Malnutrition Universal Screening Tool - MUST).
  Percentage of body fat:
  * Description: The percentage of body fat will be estimated from four skinfolds using a validated equation.
  * Unit of measurement: %
  * Interpretation: Higher percentages indicate greater adiposity.
Malnutrition Universal Screening Tool (MUST) score | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Body composition is assessed by weight (kg), height (cm), Body Mass Index (BMI = weight/height in meters squared), waist circumference, measurement of the four skinfolds (validated measurement for assessing adiposity: % body fat) and malnutrition screening (Malnutrition Universal Screening Tool - MUST).
  Risk of malnutrition (MUST) The risk of malnutrition will be assessed using the Malnutrition Universal Screening Tool (MUST). The total MUST score ranges from 0 to ≥ 2, with higher scores indicating an increased risk of malnutrition (0 = low risk; 1 = intermediate risk; ≥ 2 = high risk).
Metabolic syndrome | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  It is defined according to international recommendations (International Diabetes Federation). Diagnosis is established when at least 3 of the following criteria are present:
  1. Abdominal obesity: waist circumference > 80cm in women
  2. Elevated triglycerides: fasting triglycerides > 1.7mmol/L or current treatment for hypertriglyceridemia
  3. Reduced HDL-cholesterol: < 1.29 mmol/L in women or current treatment to increase HDL-cholesterol
  4. Elevated blood pressure: systolic blood pressure ≥ 130mmHg and/or diastolic blood pressure ≥ 85mmHg or current antihypertensive treatment
  5. Elevated fasting glucose: fasting plasma glucose ≥ 5.6mmol/L according to ADA criteria, (Note: older definitions used a threshold of ≥ 6.1mmol/L) or current treatment for type 2 diabetes or hyperglycemia
  HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) index is used to estimate insulin resistance, a key underlying mechanism of metabolic syndrome and an early marker of impaired glucose metabolism
Heart rate variability | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Heart rate is measured by ECG (Electrocardiogram) Holter over the night period at T0 and T2
GIRERD score | T2 (6 months after initiation of the Aromatase Inhibitors)
  GIRERD questionnaire is used to evaluate therapeutic adherence of patient to the Aromatase Inhibitors.
  GIRERD score; 0-6; higher score = poorer adherence
Adverse events related to the intervention | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Assessment of the occurrence of adverse events secondary to the intervention at T1 (only for the experimental group), TAPA and T2
Percentage of patients who completed all stages of the study | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  The contextual factors influencing the implementation of the APA program in real-world oncology care are evaluated using the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) framework. All 5 RE-AIM dimensions will be examined to capture key factors influencing real-world applicability, using a combination of quantitative and qualitative data collected from participants and healthcare professionals
  The first RE-AIM dimension is represented by the proportion and representativeness of individuals in the target population who participated in the intervention evaluated by percentage of patients who completed all stages of the study, dropout rate at each key stage of the study, reasons for dropout
Proportion of healthcare professionals involved in the delivery of the APA program | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  The contextual factors influencing the implementation of the APA program in real-world oncology care are evaluated using the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) framework. All 5 RE-AIM dimensions will be examined to capture key factors influencing real-world applicability, using a combination of quantitative and qualitative data collected from participants and healthcare professionals
  The third RE-AIM dimension is represented by Adoption evaluated by the engagement of individual healthcare professionals in delivering the intervention: proportion of healthcare professionals involved in the delivery of the APA program, by specialty, relative to the total number of eligible professionals at each participating site
Average number of Adapted Physical Activity (APA) sessions per week | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Fidelity of intervention is evaluated by the average number of APA sessions per week recorded throughout the intervention period using the electronic medical record.
  Unit of measure: sessions per week. Interpretation: higher values indicate greater adherence and fidelity to the intervention.
Intensity level of Physical Activity (PA) session | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Fidelity of intervention is evaluated by the intensity level of PA sessions measured by a perceived exertion scale (Borg Rating of Perceived Exertion (RPE) scale) and objective data Unit of measure: Borg RPE scale score. Higher scores indicate higher exercise intensity.
Average duration of Adapted Physical Activity (APA) sessions | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Fidelity of intervention is evaluated by the average duration of APA sessions is recorded during the intervention period using the electronic medical record.
  Unit of measurement: minutes per session. The higher the value, the longer the session.
Proportion of sessions complying with the type of exercise recommended by guidelines | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Fidelity of intervention is evaluated by proportion of sessions complying with the type of exercise recommended by guidelines.
  Unit of measure: percentage (%). Higher values indicate greater fidelity.
Program-level adaptations made during the implementation of the Adapted Physical Activity (APA) intervention | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Fidelity of intervention is evaluated by program-level adaptations made during the implementation of the APA intervention.
  This outcome is descriptive and qualitative.
Motivation scale towards health-oriented physical activity (EMAPS) total score | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Fidelity of intervention is evaluated by motivation toward APA assessed using the motivation scale towards health-oriented physical activity (EMAPS).
  Unit of measure: EMAPS total score. Interpretation: higher scores indicate higher motivation toward APA.
Patient satisfaction with the proposed Adapted Physical Activity (APA) program | From the initial phase to 6 months after the introduction of Aromatase Inhibitors.
  Fidelity of intervention is evaluated by patient satisfaction with the proposed APA program assessed using a self-administered Likert scale.
  Unit of measure: Likert scale score from 0 to 10 Interpretation: higher scores indicate greater satisfaction with the APA program.
Type of Physical Activity performed after the supervised Adapted Physical Activity (APA) program period | 6 months after the introduction of Aromatase Inhibitors
  Sustainability of PA behavior after the APA intervention is assessed at the individual level using a daily PA logbook completed by participants beyond the supervised APA program period.
  The logbook collects the following parameters daily:
  * Type of PA performed (e.g., walking, cycling, strengthening, flexibility exercises)
  * Intensity of PA, assessed using the Borg Rating of Perceived Exertion scale
  * Duration of PA expressed in minutes per session
  * Frequency of PA defined as the number of PA sessions per day and per week.
  Interpretation: higher frequency, longer duration, and higher perceived intensity of PA indicate greater sustainability of behavior change.
Intensité of Physical Activity performed after the supervised Adapted Physical Activity (APA) program period | 6 months after the introduction of Aromatase Inhibitors
  Sustainability of PA behavior after the APA intervention is assessed at the individual level using a daily PA logbook completed by participants beyond the supervised APA program period.
  The logbook collects the following parameters daily:
  * Intensity of PA, assessed using the Borg Rating of Perceived Exertion scale (Unit of measure: Borg RPE scale score.Higher scores indicate higher exercise intensity)
  * Type of PA performed (e.g., walking, cycling, strengthening, flexibility exercises)
  * Duration of PA expressed in minutes per session
  * Frequency of PA defined as the number of PA sessions per day and per week.
  Interpretation: higher frequency, longer duration, and higher perceived intensity of PA indicate greater sustainability of behavior change.
Duration of Physical Activity (PA) performed after the supervised Adapted Physical Activity (APA) program period | 6 months after the introduction of Aromatase Inhibitors
  Sustainability of PA behavior after the APA intervention is assessed at the individual level using a daily PA logbook completed by participants beyond the supervised APA program period.
  The logbook collects the following parameters daily:
  * Duration of PA expressed in minutes per session
  * Type of PA performed (e.g., walking, cycling, strengthening, flexibility exercises)
  * Intensity of PA, assessed using the Borg Rating of Perceived Exertion scale
  * Frequency of PA defined as the number of PA sessions per day and per week.
  Interpretation: higher frequency, longer duration, and higher perceived intensity of PA indicate greater sustainability of behavior change.
Frequency of Physical Activity performed after the supervised Adapted Physical Activity (APA) program period | 6 months after the introduction of Aromatase Inhibitors
  Sustainability of PA behavior after the APA intervention is assessed at the individual level using a daily PA logbook completed by participants beyond the supervised APA program period.
  The logbook collects the following parameters daily:
  * Frequency of PA defined as the number of PA sessions per day and per week.
  * Type of PA performed (e.g., walking, cycling, strengthening, flexibility exercises)
  * Intensity of PA, assessed using the Borg Rating of Perceived Exertion scale
  * Duration of PA expressed in minutes per session
  Interpretation: higher frequency, longer duration, and higher perceived intensity of PA indicate greater sustainability of behavior change.
Barriers to the long-term integration of Physical Activity (PA) into daily life and clinical practice | 6 months after the introduction of Aromatase Inhibitors
  Barriers to the long-term integration of PA into daily life and clinical practice are explored using data collected as part of the qualitative study, through semi-structured interviews conducted with patients at T2 (6 months after initiation of the Aromatase Inhibitors) and with healthcare professionals.
Facilitators to the long-term integration of Physical Activity (PA) into daily life and clinical practice | 6 months after the introduction of Aromatase Inhibitors
  Facilitators to the long-term integration of PA into daily life and clinical practice are explored using data collected as part of the qualitative study, through semi-structured interviews conducted with patients at T2 (6 months after initiation of the Aromatase Inhibitors) and with healthcare professionals.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service de Gynécologie-Obstétrique, Groupement Hospitalier Nord, Hospices Civils de Lyon, Lyon
  - Service de Chirurgie Gynécologie-Obstétrique,CHU Hôpital Nord, Saint-Priest-en-Jarez